CLINICAL TRIAL: NCT02687308
Title: Open Retropubic Radical Prostatectomy With Anterograde Anatomical Dissection Technique (RRP2A), Compared With Walsh Open Anatomical Retrograde Radical Prostatectomy (RRP)
Brief Title: Open Anterograde Radical Prostatectomy Compared to Open Retrograde Technique
Acronym: RRP2A
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Rio de Janeiro State University (Other)
Responsible Party: Principal Investigator, Fabricio Borges Carrerette, Professor, Rio de Janeiro State University
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: 41908815.9.0000.5259
Record Dates: First submitted 2015-12-22; First posted 2016-02-22 (Estimated); Last update posted 2019-04-30 (Actual); Status verified 2019-04

CONDITIONS: Prostatic Cancer; Prostatic Neoplasm
Keywords: Prostatic cancer; Radical prostatectomy; Minimally invasive prostate cancer surgery
MeSH Terms: conditions — Prostatic Neoplasms

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes

ARMS (2):
- 1Retrograde radical prostatectomy RRP (Active Comparator): This opem surgical prostatectomy techniques described by Patrick Walsh is made through prostatic dissection, from apex to the bladder neck, so the retrograde direction, the posterior layer of Denonvilliers' fascia is always included with the specimen, and urethrovesical anastomosis usually performed with multifilament interrupted suture
  Interventions: Procedure: 1 Retrograde radical prostatectomy RRP
- 2Anterograde radical prostatectomy RRP2A (Experimental): This opem surgical prostatectomy techniques dissect the prostate, bladder neck and the neurovascular bundle, in an antegrade way, from bladder neck to the apex. With careful bladder neck dissection and preservation, careful nervesparing procedures with meticulous retroprostatic dissection of the posterior layer of Denonvilliers' fascia, and urethrovesical anastomosis performed through a monofilament running suture.
  Interventions: Procedure: 2 Anterograde radical prostatectomy RRP2A

INTERVENTIONS:
Procedure: 1 Retrograde radical prostatectomy RRP — This open surgical technique described by Patrick Walsh involves prostatic dissection made from prostatic apex to the bladder neck, so the retrograde direction, the posterior layer of Denonvilliers' fascia is always included with the specimen, and urethrovesical anastomosis usually performed with multifilament interrupted suture
  Other Names: Open retrograde radical retropubic prostatectomy (RRP)
  Arms: 1Retrograde radical prostatectomy RRP
Procedure: 2 Anterograde radical prostatectomy RRP2A — This open surgical techniques performing radical retropubic prostatectomy using the same technique of minimally invasive surgery, antegrade way, from bladder neck to the apex, with careful bladder neck dissection and preservation, incremental or not careful nervesparing procedures and urethrovesical anastomosis performed by monofilament running suture, described by the Pasadena consensus for the procedure assisted by robot.
  Other Names: Open anterograde radical retropubic prostatectomy (RRP2A)
  Arms: 2Anterograde radical prostatectomy RRP2A

SUMMARY:
Prospective randomized study performing open anterograde anatomical radical retropubic prostatectomy (RRP2A) using the same technique of minimally invasive surgery described by the Pasadena consensus for the procedure assisted by robot, compared with the anatomical radical prostatectomy technique described by Patrick Walsh (RRP). Recent studies have shown benefits in the minimally invasive surgical techniques approaches, laparoscopic radical prostatectomy (LRP) and, more recently, robot-assisted radical prostatectomy (RARP). These minimally invasive techniques were associated with advantages in complications, like intraoperative bleeding, transfusion rates and in earlier recovery of important genitourinary functions such as urinary continence and penile erection. But still has not been demonstrated conclusively advantages as oncological control and it is believed that there are about 200 to 250 cases of learning curve so that the rates of complications and positive surgical margins become stable and similar to the open radical prostatectomy. These facts associated with the high cost of robotic technology still have limited the generalization of this approach in many developing countries such as Brazil. While the majority of studies made by comparing the radical prostatectomy (RP), robot X laparoscopic X open, show a slight advantage in the first two, there is a significant bias in these studies, which is that the surgical technique used in each procedure differs significantly from minimally invasive and open surgical techniques. The evolution of minimally invasive radical prostatectomy was based on an entirely different anatomical benchmark of that described by Patrick Walsh. While robotics and laparoscopic techniques dissect the prostate, bladder neck and the neurovascular bundle in an antegrade way, from bladder neck to the apex, the Walsh RRP technique is completely different in several ways, the dissection is made from prostatic apex to the bladder neck, so the retrograde direction, the posterior layer of Denonvilliers' fascia, is always included with the specimen, and urethrovesical anastomosis, usually performed with multifilament interrupted suture, only for indicating the major differences. The RRP2A will be performed by incision (open surgery) and will be compared with the anatomical radical prostatectomy technique described by Patrick Walsh RRP, and performed by the same surgeons.

DETAILED DESCRIPTION:
Introduction The best way to treat localized prostate cancer is radical prostatectomy (RP). This surgery has been performed since 1905, introduced by Young. Initial results were disappointing due to high rates of bleeding, incontinence, impotence and other surgical complications. It was from the knowledge of the anatomical basis of vascularization and innervation of male pelvis by Patrick Walsh that the radical retropubic prostatectomy (RRP) had its development and has become the first choice in the treatment of initial stages of prostate cancer.

Large series of literature results show excellent long-term cancer control, with about 80% of patients with no evidence of disease (biochemical or clinical) in 10 years.

Urinary incontinence rates after RRP vary widely, those regarding absence of the urinary incontinence after 18 months of surgery are uniform in presenting continence rates above 90%. However the continence rates over the short term are much lower.

The definition of recovery of sexual function after surgery is the ability to keep satisfactory sexual intercourse with or without the use of oral drugs. The key factors for the recovery of erectile capacity power prior to surgery are the patient's age and the surgical technique employed. Academic series of open RRP report recovery rates of about 70% with bilateral preservation of nerves, and about 50% with unilateral preservation after 18 months.

Recent studies have shown benefits in the minimally invasive approaches, laparoscopic radical prostatectomy (LRP) and, more recently, robot-assisted radical prostatectomy (RARP), with respect to complications like intraoperative bleeding, but still do not demonstrate conclusively advantages as oncological control. However the recovery of erectile function and urinary continence seems to recover better and earlier. It is believed that there are about 200-250 cases of learning curve to reach levels that the rates of complications and positive surgical margins become stable and similar to the open radical prostatectomy, and the high cost of robotic technology still has limited the generalization of this approach in many countries.

The exponential adoption of minimally invasive robot-assisted radical prostatectomy (RARP) has been remarkable and unprecedented. According to unverified estimates from the Da Vinci surgical system manufacturer (Intuitive Surgical, Sunnyvale, CA) over 80% of radical prostatectomy within the US were performed robotically in 2010. This dramatic shift in radical prostatectomy practice patterns occurred despite the lack of evidence of high quality of the method, not yet demonstrating its oncology benefits, safety or cost effectiveness compared to open surgery.

While the majority of studies made by comparing the radical prostatectomy: robot X laparoscopic X open, show a slight advantage in the first two in regard intraoperative complications, especially bleeding, and post operative complications as the speed of recovery of continence and sexual potency. There is a significant bias in these studies, which is that the surgical technique used in each procedure differs significantly from minimally invasive and open surgical techniques. The evolution of minimally invasive prostate surgery was based on an entirely different anatomical benchmark of that described by Patrick Walsh for open radical prostatectomy.

While robotics and laparoscopic techniques dissect the prostate, bladder neck and the neurovascular bundle, in an antegrade way, from bladder neck to the apex. With careful bladder neck dissection and preservation, incremental or not careful nerve-sparing procedures with meticulous rectoprostatic dissection of the posterior layer of Denonvilliers' fascia, with the aim of maximizing the preservation of the fibers located within the periprostatic tissue that covers the lateral and anterior surface of the prostate, and urethrovesical anastomosis performed through a monofilament running suture. The Walsh open radical retropubic prostatectomy (RRP) technique is completely different in several ways, the dissection is made from prostatic apex to the bladder neck, so the retrograde direction, the posterior layer of Denonvilliers' fascia is always included with the specimen, and urethrovesical anastomosis usually performed with multifilament interrupted suture, only for indicating the major differences.

This trial proposes a prospective randomized study performing radical prostatectomy due to open surgery using the same technique of minimally invasive surgery, antegrade, from bladder neck to the apex, with careful bladder neck dissection and preservation, incremental or not careful nerve-sparing procedures and urethrovesical anastomosis performed by monofilament running suture, described by the Pasadena consensus for the procedure assisted by robot.

A pilot study was performed to test the feasibility of this technique and managed to complete ten surgeries in all its stages without conversion to the standard radical prostatectomy technique of Patrick Walsh.

Patients and methods

This technique will be performed by incision (open surgery) and will be compared with the anatomical radical prostatectomy technique described by Patrick Walsh and performed by the same surgeons.

Two hundred and forty patients will be selected with localized prostate cancer with indication for radical surgery, confirmed by biopsy and staged as protocol of urology service HUPE UERJ of Rio de Janeiro, Brazil.

Patients will be randomized into two arms, according to the kind of technique, and in three sets according to the three different main surgeons. Randomization was performed by software on the site "www.randomizer.org/" on November 17, 2015, as follows:

Arm 1 - open retrograde radical retropubic prostatectomy (RRP).

Arm 2 - open anterograde anatomical radical retropubic prostatectomy (RRP2A).

Set 1 - Surgeon A. 1, 1, 2, 2, 1, 2, 2, 2, 1, 1, 1, 2, 1, 1, 1, 2, 2, 1, 1, 1, 1, 2, 2, 1, 2, 2, 1, 2, 1, 2, 2, 2, 2, 2, 2, 1, 2, 1, 1, 2, 2, 2, 1, 1, 2, 2, 2, 2, 2, 2, 2, 1, 2, 1, 2, 2, 1, 1, 2, 2, 1, 2, 1, 2, 1, 1, 2, 2, 2, 2, 1, 1, 1, 1, 2, 1, 1, 1, 1, 1

Set 2 - Surgeon B. 2, 2, 2, 1, 1, 2, 1, 1, 1, 2, 1, 1, 1, 2, 1, 2, 2, 2, 2, 1, 1, 2, 2, 2, 2, 2, 2, 2, 2, 1, 1, 2, 2, 2, 1, 2, 2, 2, 2, 2, 2, 1, 2, 2, 1, 2, 1, 2, 1, 1, 1, 2, 2, 2, 1, 2, 2, 2, 2, 1, 2, 2, 2, 2, 1, 1, 2, 2, 2, 2, 2, 1, 1, 2, 2, 2, 1, 2, 2, 1

Set 3 - Surgeon C. 2, 2, 1, 2, 2, 1, 1, 1, 1, 1, 2, 2, 2, 2, 1, 2, 2, 1, 2, 2, 1, 1, 1, 2, 2, 1, 2, 1, 2, 2, 2, 2, 2, 1, 1, 1, 2, 2, 2, 1, 2, 1, 1, 2, 1, 2, 1, 1, 1, 2, 1, 2, 1, 1, 1, 2, 2, 1, 1, 1, 1, 2, 2, 1, 1, 1, 2, 2, 2, 1, 1, 1, 1, 1, 1, 2, 2, 1, 2, 2

A prostatectomy technique of "open anterograde anatomical radical retropubic prostatectomy (RRP2A)" dissects the prostate, bladder neck and the neurovascular bundle, antegrade, from bladder neck to the apex, with careful bladder neck dissection and preservation, incremental or not careful nerve-sparing procedures with meticulous rectoprostatic dissection of the posterior layer of Denonvilliers' fascia, with the aim of maximizing the preservation of the fibers located within the periprostatic tissue that covers the lateral and anterior surface of the prostate, and urethrovesical anastomosis performed through a monofilament running suture, follow the step-by-step described in Pasadena consensus for robot-assisted radical prostatectomy and adapted to open surgery.

Selection of Study Population Patients will be selected with localized prostate cancer confirmed by biopsy and staged as protocol of urology service of Pedro Ernesto Hospital of State University of Rio de Janeiro, Brazil (HUPE UERJ). All patients with localized prostate cancer and indication for open radical retropubic prostatectomy (RRP) will be invited to participate in this study.

The Visits Procedures:

Day 0. Screening may be performed before or in the same visit of Randomization with the patient signed the informed consent before or in the day of surgery.

Evaluation of inclusion and exclusion criteria. Randomization may also be performed just before starting the surgical procedure. Patient identification as age and race, as well data as result of the biopsy, prostate specific antigen (PSA) levels and clinical stage are transcribed to the protocol. The surgery information is recorded in details at the end of surgery. Model protocol annotation form in appendix 1.

Visit 1 - Day 7 to RRP2A and day 14 for RRP. In this visit the bladder catheter is taken and collected information of postoperative complications, time and drainage volume of suction drain, wound aspect, length of hospital stay.

After removal of the bladder catheter will be observed if the patient has a urethral drip or if he can retain urine in the bladder.

PSA dosage will be requested. Visit 2 - Day 30. This visit will be harvested postoperative complications information, PSA results and the result of the pathological examination of the surgical specimens, prostate, seminal vesicles and pelvic nodes. Evaluation of the surgical margins, urethral, bladder and circumferential and pathological staging.

In this visit will be applied two questionnaires for evaluation of urinary continence and sexual function, International Consultation on Incontinence Questionnaire - Short Form (ICIQ-SF) and International Index of Erectile Function-5 (IIEF5).

In this visit the patients will also be asked about their continence, if they are completely continent, ie, without the use of any pad, or partial continent, use of only one pad per day for protection against accidents. If this one pad is used only to protect any occasional urine leakage, but not wets every day, he will be asked how many times a week this pad is wet, with the following response options: once, twice, three times or more, almost every day or all days of the week. If the patient answers that the pad wets once or twice a week, he will be considered partial continent, to answer it wets three or more times, almost every day or every day of the week, the patient will be considered incontinent.

Visit 3 - Day 60. This visit will be harvested postoperative complications information, PSA results and the result of the pathological examination of the surgical specimens if these results are not ready in the previous visit. Application of the questionnaires ICIQ-SF and IIEF5. In this visit will also be asked to the patients about their continence, classified as completely continent, partial continent and incontinent. They will be also asked about sexual intercourse with penetration and if they are using medication as phosphodiesterase type 5 (PDE5) inhibitors.

Visit 4 - Day 90. This visit will be harvested postoperative complications information and PSA results.

Application of the questionnaires ICIQ-SF and IIEF5. In this visit it will also be asked to the patients about their continence, classified as completely continent, partial continent and incontinent. They will be ask also about sexual intercourse with penetration and if they are using medication as PDE5 inhibitors.

Visit 5 - Day 180. This visit will be assessed the result of PSA. Application of the questionnaires ICIQ-SF and IIEF5 and asked to patients about their continence, classified as completely continent, partial continent and incontinent. They will also be asked about sexual intercourse with penetration and if they are using medication as PDE5 inhibitors.

Visit 6 - 1 year - End of Study. This visit will be assessed the result of PSA. Application of the questionnaires ICIQ-SF and IIEF5 and ask the patients about their continence, classified as completely continent, partial continent and incontinent. They will also be asked about sexual intercourse with penetration and if they are using medication as PDE5 inhibitors.

ELIGIBILITY:
Inclusion Criteria:

1. Age 40 years or older and willing and able to provide informed consent;
2. Histologically and clinically confirmed localized adenocarcinoma of the prostate without neuroendocrine differentiation, signet cell, or small cell features;
3. Surgical indication for open radical prostatectomy;
4. PSA less than 20 ng/mL;
5. No evidence of metastasis disease;
6. Cleared by the primary medical doctor for surgery;
7. No prior systemic therapy for prostate cancer;
8. Eastern Cooperative Oncology Group (ECOG) performance status of 0 or 1.

Exclusion Criteria:

1. Refuses to give informed consent;
2. Refuses or is unable to have radical prostatectomy;
3. Stage T4;
4. Deemed a poor surgical risk per primary medical doctor;
5. Received prior therapeutic intervention for prostate cancer;
6. Deep vein thrombosis (DVT)/pulmonary embolism (PE) in the past 6 months;
7. Neurogenic bladder;
8. Urinary incontinence.

Ages: 40 Years to 80 Years | Sex: Male | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 240 (Actual)
Dates: Start 2016-03; Primary Completion 2019-04 (Actual); Study Completion 2019-04 (Actual)

PRIMARY OUTCOMES:
Surgical time for completed prostatectomy | Day of surgery
  Measurement of time for completed surgery. The median operative duration will be measured in minutes and compared between the two techniques

SECONDARY OUTCOMES:
PSA | One year
  The rate of patients who have an undetectable PSA after surgery
Time of urinary catheter | Three months
  Time of catheter removal
Time of urethrovesical anastomosis | Day of surgery
  Time to accomplish urethrovesical anastomosis. The median duration of urethrovesical anastomosis will be measured in minutes and compared between the two techniques
Hospital length of stay | One month
  Measurement of hospital stay
Positive surgical margins | Three months
  The rate of patients who have an positive surgical margins
Urinary Continence | One year
  The rate of patients who have complete recovery of urinary continence. At the time of catheter removal all patients who have a dry safety pad within the first 24 h will be define as continent. Urinary continence will be evaluate using the International Consultation of Incontinence Questionnaire of Urinary Incontinence (ICIQ-UI) short-form instrument.
Erectile function | One year
  The rate of patients who have complete recovery of erectile function. Erectile function will be evaluate using the International Index of Erectile Function (IIEF-5)
Surgical complication | Three months postsurgery
  Accurate reporting based on the classification of Clavien-Dindo system such as lymphorrhea, lymphocele, bleeding, perioperative transfusion rate, pelvic hematoma, urine leakage and disrupted anastomosis.
Postoperative complications | One year
  Accurate reporting of postoperative complications such as bladder neck contractures

CONTACTS AND LOCATIONS:
Overall Officials: Fabricio B Carrerette, Principal Investigator — State University of Rio de Janeiro
Locations (1):
- State University of Rio de Janeiro, Rio de Janeiro, Brazil

IPD SHARING:
Plan to Share IPD: Yes
through a table without identifying the name but with the initial and the registration number in the institution
Supporting Information: Study Protocol, SAP, ICF, CSR
Time Frame: The study will be alowed when statistical analyses data and results are completed after article is published and estimated time for one year.
Access Criteria: Men diagnosed with localized prostatic cancer and indication of radical prostatectomy. Exclusion criteria: clinical contra indications for surgery, local advanced prostate cancer and PSA marker up to 20 ng/dL.

REFERENCES:
- [Background] Yatani R, Chigusa I, Akazaki K, Stemmermann GN, Welsh RA, Correa P. Geographic pathology of latent prostatic carcinoma. Int J Cancer. 1982 Jun 15;29(6):611-6. doi: 10.1002/ijc.2910290602. PMID 7107064
- [Background] Ficarra V, Borghesi M, Suardi N, De Naeyer G, Novara G, Schatteman P, De Groote R, Carpentier P, Mottrie A. Long-term evaluation of survival, continence and potency (SCP) outcomes after robot-assisted radical prostatectomy (RARP). BJU Int. 2013 Aug;112(3):338-45. doi: 10.1111/bju.12001. Epub 2013 Mar 7. PMID 23470027
- [Result] Walsh PC, Donker PJ. Impotence following radical prostatectomy: insight into etiology and prevention. J Urol. 1982 Sep;128(3):492-7. doi: 10.1016/s0022-5347(17)53012-8. No abstract available. PMID 7120554
- [Result] Mohler J, Bahnson RR, Boston B, Busby JE, D'Amico A, Eastham JA, Enke CA, George D, Horwitz EM, Huben RP, Kantoff P, Kawachi M, Kuettel M, Lange PH, Macvicar G, Plimack ER, Pow-Sang JM, Roach M 3rd, Rohren E, Roth BJ, Shrieve DC, Smith MR, Srinivas S, Twardowski P, Walsh PC. NCCN clinical practice guidelines in oncology: prostate cancer. J Natl Compr Canc Netw. 2010 Feb;8(2):162-200. doi: 10.6004/jnccn.2010.0012. No abstract available. PMID 20141676
- [Result] Walsh PC, Partin AW, Epstein JI. Cancer control and quality of life following anatomical radical retropubic prostatectomy: results at 10 years. J Urol. 1994 Nov;152(5 Pt 2):1831-6. doi: 10.1016/s0022-5347(17)32396-0. PMID 7523730
- [Result] Eastham JA, Scardino PT, Kattan MW. Predicting an optimal outcome after radical prostatectomy: the trifecta nomogram. J Urol. 2008 Jun;179(6):2207-10; discussion 2210-1. doi: 10.1016/j.juro.2008.01.106. Epub 2008 Apr 18. PMID 18423693
- [Result] Catalona WJ, Carvalhal GF, Mager DE, Smith DS. Potency, continence and complication rates in 1,870 consecutive radical retropubic prostatectomies. J Urol. 1999 Aug;162(2):433-8. PMID 10411052
- [Result] Kundu SD, Roehl KA, Eggener SE, Antenor JA, Han M, Catalona WJ. Potency, continence and complications in 3,477 consecutive radical retropubic prostatectomies. J Urol. 2004 Dec;172(6 Pt 1):2227-31. doi: 10.1097/01.ju.0000145222.94455.73. PMID 15538237
- [Result] Bolenz C, Gupta A, Hotze T, Ho R, Cadeddu JA, Roehrborn CG, Lotan Y. Cost comparison of robotic, laparoscopic, and open radical prostatectomy for prostate cancer. Eur Urol. 2010 Mar;57(3):453-8. doi: 10.1016/j.eururo.2009.11.008. Epub 2009 Nov 11. PMID 19931979
- [Result] Secin FP, Savage C, Abbou C, de La Taille A, Salomon L, Rassweiler J, Hruza M, Rozet F, Cathelineau X, Janetschek G, Nassar F, Turk I, Vanni AJ, Gill IS, Koenig P, Kaouk JH, Martinez Pineiro L, Pansadoro V, Emiliozzi P, Bjartell A, Jiborn T, Eden C, Richards AJ, Van Velthoven R, Stolzenburg JU, Rabenalt R, Su LM, Pavlovich CP, Levinson AW, Touijer KA, Vickers A, Guillonneau B. The learning curve for laparoscopic radical prostatectomy: an international multicenter study. J Urol. 2010 Dec;184(6):2291-6. doi: 10.1016/j.juro.2010.08.003. Epub 2010 Oct 16. PMID 20952022
- [Result] Lowrance WT, Tarin TV, Shariat SF. Evidence-based comparison of robotic and open radical prostatectomy. ScientificWorldJournal. 2010 Nov 16;10:2228-37. doi: 10.1100/tsw.2010.218. PMID 21103791
- [Result] Binder J, Kramer W. Robotically-assisted laparoscopic radical prostatectomy. BJU Int. 2001 Mar;87(4):408-10. doi: 10.1046/j.1464-410x.2001.00115.x. No abstract available. PMID 11251539
- [Result] Menon M, Shrivastava A, Tewari A, Sarle R, Hemal A, Peabody JO, Vallancien G. Laparoscopic and robot assisted radical prostatectomy: establishment of a structured program and preliminary analysis of outcomes. J Urol. 2002 Sep;168(3):945-9. doi: 10.1016/S0022-5347(05)64548-X. PMID 12187196
- [Result] Montorsi F, Wilson TG, Rosen RC, Ahlering TE, Artibani W, Carroll PR, Costello A, Eastham JA, Ficarra V, Guazzoni G, Menon M, Novara G, Patel VR, Stolzenburg JU, Van der Poel H, Van Poppel H, Mottrie A; Pasadena Consensus Panel. Best practices in robot-assisted radical prostatectomy: recommendations of the Pasadena Consensus Panel. Eur Urol. 2012 Sep;62(3):368-81. doi: 10.1016/j.eururo.2012.05.057. Epub 2012 Jun 7. PMID 22763081
- [Result] Sciarra A, Cristini C, Von Heland M, Salciccia S, Gentile V. Randomized trial comparing an anterograde versus a retrograde approach to open radical prostatectomy: results in terms of positive margin rate. Can Urol Assoc J. 2010 Jun;4(3):192-8. doi: 10.5489/cuaj.09089. PMID 20514284
- [Result] Pierorazio PM, Mullins JK, Eifler JB, Voth K, Hyams ES, Han M, Pavlovich CP, Bivalacqua TJ, Partin AW, Allaf ME, Schaeffer EM. Contemporaneous comparison of open vs minimally-invasive radical prostatectomy for high-risk prostate cancer. BJU Int. 2013 Oct;112(6):751-7. doi: 10.1111/j.1464-410X.2012.11757.x. Epub 2013 Jan 28. PMID 23356390
- [Result] Ficarra V, Novara G, Mottrie A, Wilson TG, Montorsi F. Reply to Robert P. Myers' letter to the editor re: Francesco Montorsi, Timothy G. Wilson, Raymond C. Rosen, et al. best practices in robot-assisted radical prostatectomy: recommendations of the Pasadena consensus panel. Eur Urol 2012;62:368-81. Eur Urol. 2013 Mar;63(3):e42-3. doi: 10.1016/j.eururo.2012.11.036. Epub 2012 Nov 22. No abstract available. PMID 23253772
- [Result] Novara G, Ficarra V, Rosen RC, Artibani W, Costello A, Eastham JA, Graefen M, Guazzoni G, Shariat SF, Stolzenburg JU, Van Poppel H, Zattoni F, Montorsi F, Mottrie A, Wilson TG. Systematic review and meta-analysis of perioperative outcomes and complications after robot-assisted radical prostatectomy. Eur Urol. 2012 Sep;62(3):431-52. doi: 10.1016/j.eururo.2012.05.044. Epub 2012 Jun 2. PMID 22749853
- [Result] Ficarra V, Novara G, Rosen RC, Artibani W, Carroll PR, Costello A, Menon M, Montorsi F, Patel VR, Stolzenburg JU, Van der Poel H, Wilson TG, Zattoni F, Mottrie A. Systematic review and meta-analysis of studies reporting urinary continence recovery after robot-assisted radical prostatectomy. Eur Urol. 2012 Sep;62(3):405-17. doi: 10.1016/j.eururo.2012.05.045. Epub 2012 Jun 1. PMID 22749852
- [Result] Novara G, Ficarra V, Mocellin S, Ahlering TE, Carroll PR, Graefen M, Guazzoni G, Menon M, Patel VR, Shariat SF, Tewari AK, Van Poppel H, Zattoni F, Montorsi F, Mottrie A, Rosen RC, Wilson TG. Systematic review and meta-analysis of studies reporting oncologic outcome after robot-assisted radical prostatectomy. Eur Urol. 2012 Sep;62(3):382-404. doi: 10.1016/j.eururo.2012.05.047. Epub 2012 Jun 2. PMID 22749851
- [Result] Ficarra V, Novara G, Ahlering TE, Costello A, Eastham JA, Graefen M, Guazzoni G, Menon M, Mottrie A, Patel VR, Van der Poel H, Rosen RC, Tewari AK, Wilson TG, Zattoni F, Montorsi F. Systematic review and meta-analysis of studies reporting potency rates after robot-assisted radical prostatectomy. Eur Urol. 2012 Sep;62(3):418-30. doi: 10.1016/j.eururo.2012.05.046. Epub 2012 Jun 1. PMID 22749850
- [Result] Novara G, Ficarra V, D'elia C, Secco S, Cioffi A, Cavalleri S, Artibani W. Evaluating urinary continence and preoperative predictors of urinary continence after robot assisted laparoscopic radical prostatectomy. J Urol. 2010 Sep;184(3):1028-33. doi: 10.1016/j.juro.2010.04.069. PMID 20643426
- [Result] Novara G, Ficarra V, D'Elia C, Secco S, Cavalleri S, Artibani W. Trifecta outcomes after robot-assisted laparoscopic radical prostatectomy. BJU Int. 2011 Jan;107(1):100-4. doi: 10.1111/j.1464-410X.2010.09505.x. PMID 20633003
- [Result] Novara G, Ficarra V, D'Elia C, Secco S, Cavalleri S, Artibani W. Prospective evaluation with standardised criteria for postoperative complications after robotic-assisted laparoscopic radical prostatectomy. Eur Urol. 2010 Mar;57(3):363-70. doi: 10.1016/j.eururo.2009.11.032. Epub 2009 Nov 21. PMID 19944519
- [Result] Ficarra V, Novara G, Secco S, D'Elia C, Boscolo-Berto R, Gardiman M, Cavalleri S, Artibani W. Predictors of positive surgical margins after laparoscopic robot assisted radical prostatectomy. J Urol. 2009 Dec;182(6):2682-8. doi: 10.1016/j.juro.2009.08.037. PMID 19836778
- [Result] Ficarra V, Novara G, Fracalanza S, D'Elia C, Secco S, Iafrate M, Cavalleri S, Artibani W. A prospective, non-randomized trial comparing robot-assisted laparoscopic and retropubic radical prostatectomy in one European institution. BJU Int. 2009 Aug;104(4):534-9. doi: 10.1111/j.1464-410X.2009.08419.x. Epub 2009 Mar 5. PMID 19281468
- [Result] Ficarra V, Novara G, Artibani W, Cestari A, Galfano A, Graefen M, Guazzoni G, Guillonneau B, Menon M, Montorsi F, Patel V, Rassweiler J, Van Poppel H. Retropubic, laparoscopic, and robot-assisted radical prostatectomy: a systematic review and cumulative analysis of comparative studies. Eur Urol. 2009 May;55(5):1037-63. doi: 10.1016/j.eururo.2009.01.036. Epub 2009 Jan 25. PMID 19185977
- [Result] Artibani W, Fracalanza S, Cavalleri S, Iafrate M, Aragona M, Novara G, Gardiman M, Ficarra V. Learning curve and preliminary experience with da Vinci-assisted laparoscopic radical prostatectomy. Urol Int. 2008;80(3):237-44. doi: 10.1159/000127333. Epub 2008 May 14. PMID 18480623
- [Result] Fracalanza S, Ficarra V, Cavalleri S, Galfano A, Novara G, Mangano A, Plebani M, Artibani W. Is robotically assisted laparoscopic radical prostatectomy less invasive than retropubic radical prostatectomy? Results from a prospective, unrandomized, comparative study. BJU Int. 2008 May;101(9):1145-9. doi: 10.1111/j.1464-410X.2008.07513.x. PMID 18399830
- [Result] Tewari A, Takenaka A, Mtui E, Horninger W, Peschel R, Bartsch G, Vaughan ED. The proximal neurovascular plate and the tri-zonal neural architecture around the prostate gland: importance in the athermal robotic technique of nerve-sparing prostatectomy. BJU Int. 2006 Aug;98(2):314-23. doi: 10.1111/j.1464-410X.2006.06266.x. PMID 16879671